CLINICAL TRIAL: NCT07007663
Title: A Single-center Observational Study Looking at the Prevalence of Directional Preference in the Lumbar Stenosis Population for Low Back Pain Patients
Brief Title: The Prevalence of Directional Preference in the Lumbar Stenosis Population
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 24-01830
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Stenosis
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumbar stenosis patients: Patients undergoing physical therapy treatment at an outpatient clinic will be enrolled. Data collection will include patient outcome measures, if directional preference is present and results from the functional tests performed by 3 licensed physical therapists who also hold their diploma in the McKenzie Method of Mechanical Diagnosis and Therapy (specialized training in recognizing directional preference) as a part of routine care (not research) for the enrolled patients. Data will be collected at initial onset, at discharge, and at a 6 months follow up.

SUMMARY:
This will be a prospective cohort observational study observing patients with low back pain with leg pain who present for outpatient physical therapy care at Rusk Rehabilitation at NYU Langone Ambulatory Care Lake Success. Patients are eligible if they present with imaging of stenosis in their lumbar spine on MRI or CT Scan and note radicular leg symptoms with associated neurological deficits on the physical examination for at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Neurogenic claudication (pain in the buttock, thigh, or leg during ambulation) or radicular leg symptoms with associated neurological deficits on the physical examination for at least 12 weeks.
* Confirmatory cross-sectional magnetic resonance imaging (MRI) or computed tomography (CT) imaging demonstrating the presence of either central or lateral lumbar spinal stenosis at one or more levels was required.
* Age >48 years old
* Willing and able to consent
* Scheduled to receive physical therapy that includes the collection of patients outcomes, functional tests, and may include the conduct of a two-stage treadmill test

Exclusion Criteria:

* Radiographic evidence of instability, degenerative spondylolisthesis, fracture, or scoliosis of more than 15°.
* Comorbid health conditions precluding surgical management, prior lumbar surgery, progressive neurological deficit, any inflammatory conditions such as rheumatoid arthritis or indication of a potential non-musculoskeletal spinal condition (e.g., active malignancy, infection, etc.)

Min Age: 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that choose to participate are undergoing a course of outpatient physical therapy care on their own accord with a referral to physical therapy. The participants have the ability to drop out or withdraw at any point of the study.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of directional preference (DP) among patients diagnosed with lumbar spinal stenosis (LSS) | Baseline
  Prevalence is calculated as the proportion of patients with DP out of the total sample of LSS patients.
Prevalence of DP among patients diagnosed with LSS | Visit 3 (variable by participant; up to Day 365)
  Prevalence is calculated as the proportion of patients with DP out of the total sample of LSS patients.

SECONDARY OUTCOMES:
Prevalence of Specific Directions of Directional Preference (DP) in LSS Population | Visit 3 (variable by participant; up to Day 365)
  Percentage of patients with LSS demonstrating each primary DP movement direction (FLEXION, EXTENSION, or LATERAL).
Change in Pain Scores in LSS Patients With and Without DP | Baseline, Visit 3 (variable by participant; up to Day 365)
  Pain is measured using the Numeric Pain Rating Scale (NPRS), a self-report scale where individuals rate their pain level on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
Change in Pain Scores in LSS Patients With and Without DP | Baseline, 6 Months Post-Visit 3 (variable by participant; up to Day 365 + 6 Months)
  Pain is measured using the Numeric Pain Rating Scale (NPRS), a self-report scale where individuals rate their pain level on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference Score in LSS Patients With and Without DP | Baseline, Visit 3 (variable by participant; up to Day 365)
  The PROMIS Pain Interference questionnaire is a 40-item measure of the extent to which pain interferes with various aspects of a person's life. Each item is rated on a Likert scale from 1-5; the raw score is the sum of item responses. The raw score is standardized into an overall T-score ranging from 0-100, with a mean of 50 and standard deviation of 10. Higher scores indicate greater pain interference.
Change in PROMIS - Pain Interference Score in LSS Patients With and Without DP | Baseline, 6 Months Post-Visit 3 (variable by participant; up to Day 365 + 6 Months)
  The PROMIS Pain Interference questionnaire is a 40-item measure of the extent to which pain interferes with various aspects of a person's life. Each item is rated on a Likert scale from 1-5; the raw score is the sum of item responses. The raw score is standardized into an overall T-score ranging from 0-100, with a mean of 50 and standard deviation of 10. Higher scores indicate greater pain interference.
Change in PROMIS - Physical Function Score in LSS Patients With and Without DP | Baseline, Visit 3 (variable by participant; up to Day 365)
  The PROMIS Physical Function questionnaire is a 165-item measure of a patient's self-reported capability to perform functional activities, including activities of daily living (ADLs) and activities in the community. Each item is rated on a Likert scale from 1-5; the raw score is the sum of item responses. The raw score is standardized into an overall T-score ranging from 0-100, with a mean of 50 and standard deviation of 10. Higher scores indicate greater physical function.
Change in PROMIS - Physical Function Score in LSS Patients With and Without DP | Baseline, 6 Months Post-Visit 3 (variable by participant; up to Day 365 + 6 Months)
  The PROMIS Physical Function questionnaire is a 165-item measure of a patient's self-reported capability to perform functional activities, including activities of daily living (ADLs) and activities in the community. Each item is rated on a Likert scale from 1-5; the raw score is the sum of item responses. The raw score is standardized into an overall T-score ranging from 0-100, with a mean of 50 and standard deviation of 10. Higher scores indicate greater physical function.

CONTACTS AND LOCATIONS:
Overall Officials: William Oswald, DPT, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No